CLINICAL TRIAL: NCT05370924
Title: Assessment and Risk Stratification of the Development of Postoperative Persistent Postoperative Pain in Patients Undergoing Orthopedic Surgery
Brief Title: Assessment of the Development of Postoperative Persistent Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Maurizio Berardino, Director, A.O.U. Città della Salute e della Scienza
Other Study IDs: DOROTHEA
Record Dates: First submitted 2022-02-02; First posted 2022-05-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use; Post Operative Pain; Chronic Pain
Keywords: postoperative pain; opioid naive; opioid tolerant; orthopedic surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the postoperative period, it is possible to observe the development of acute pain, which lasts no longer than a week after surgery. However, sometimes some patients see the prolongation of this pain beyond the healing time of the tissue, turning into a chronic condition. Persistent postoperative pain is a disease with a complex and still unknown etiology, affecting between 5 and 75% of the population. The development of persistent postoperative pain is a rather important issue since the physician managing the patient must on the one hand ensure adequate analgesia, and on the other hand, minimize the risk of continued opioid use in the case of chronicization.

In a study conducted analyzing the prevalence of persistent postoperative pain in various surgeries it was seen to occur more frequently in limb amputation (prevalence >85%), thoracotomy (prevalence 48%), knee arthroplasty (prevalence 44%), laminectomies, and spinal arthrodesis (prevalence 5-46%), and hip replacement (prevalence 27%) making this type of pain more frequent in the patient undergoing orthopedic surgery.

As the mechanisms behind its development have not yet been fully clarified, efforts to study the clinical factors associated with the onset of this pathology have been attempted.

As there is no way in the literature to stratify the risk of the population in order to prevent the development of postoperative pain, based on the variables reported by different studies, it was decided to administer in patients referred to the Orthopedics and Traumatology 1 U and Orthopedics and Traumatology 3 U department at the Orthopedic Trauma Center of Turin questionnaires to assess the development of chronic pain for screening purposes and to contribute to the improvement of the long-term management of these patients in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthopedic surgery considered at high risk of developing persistent postoperative pain (i.e. knee prothesic surgery, hip prothesic surgery, spine fusion surgery)

Exclusion Criteria:

* Patients undergoing redo prothesic surgery
* Trauma patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing orthopedic surgery considered at high risk of developing persistent postoperative pain (i.e. knee prothesic surgery, hip prothesic surgery, spine fusion surgery)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Persistent and chronic postsurgical pain | 48 hrs, 2 weeks, 3 months
  Presence or not of posturgical pain, persistent NRS > 4 in surgical area

SECONDARY OUTCOMES:
NRS | 3 months
  pain
Postsurgical complications | 3 months
  Presence y/n of surgical complications
Anxiety | 3 months
  Psychometric test, GAD-7
Depression | 3 months
  Psychometric test, PHQ-9

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio ospedaliero CTO, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steyaert A, Lavand'homme P. Prevention and Treatment of Chronic Postsurgical Pain: A Narrative Review. Drugs. 2018 Mar;78(3):339-354. doi: 10.1007/s40265-018-0866-x. PMID 29380289
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Tiippana E, Hamunen K, Heiskanen T, Nieminen T, Kalso E, Kontinen VK. New approach for treatment of prolonged postoperative pain: APS Out-Patient Clinic. Scand J Pain. 2016 Jul;12:19-24. doi: 10.1016/j.sjpain.2016.02.008. Epub 2016 Mar 11. PMID 28850486